CLINICAL TRIAL: NCT04200053
Title: The Effect of Reflexology Massage and Passive Music Therapy Intervention Before Burn Dressing on Pain, Anxiety Level and Sleep Quality
Brief Title: The Effect of Reflexology Massage and Passive Music Therapy Intervention Before Burn Dressing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Ayse Kabuk, RN, PhD, Research Assistant, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Record Dates: First submitted 2019-11-21; First posted 2019-12-16 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Burn Degree Second; Burn Degree Third
Keywords: burn; reflexology; music; pain; anxiety; sleep
MeSH Terms: conditions — Burns; Pain; Anxiety Disorders | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Intervention Model Description: Grup 1: Reflexology massage group Grup 2: Reflexology massage and pasiive music group Grup 3: Control group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Reflexology massage (Experimental): Reflexology massage
  Interventions: Other: Reflexology massage
- Reflexology massage and passive music (Experimental): Reflexology massage and passive music
  Interventions: Other: Reflexology massage and passive music
- Control (No Intervention): Control

INTERVENTIONS:
Other: Reflexology massage — Before the burn dressing, a reflexology massage will be performed for 20 minutes on the right foot and 20 minutes on the left foot. This intervention will continue in the morning for 3 days.
  Arms: Reflexology massage
Other: Reflexology massage and passive music — Before the burn dressing, a reflexology massage and passive music will be performed for 20 minutes on the right foot and 20 minutes on the left foot. Instrumental music will be played during the massage. This intervention will continue in the morning for 3 days.
  Arms: Reflexology massage and passive music

SUMMARY:
Reflexology massage applied before burn dressing reduces pain, anxiety and sleep problems

DETAILED DESCRIPTION:
Reflexology massage regulates blood circulation and energy, gives a feeling of relaxation and provides homeostasis. During reflexology massage, relaxation music is recommended because it contributes to the relaxation of the individual. In the literature, reflexology massage and music therapy are used in different pain management, and these methods reduce anxiety and improve sleep quality. However, there is no study in which reflexology massage and passive music therapy are used to reduce pain, anxiety and sleep problems associated with dressing of burn individuals. It is thought that reflexology massage and passive music therapy will reduce pain, anxiety and sleep problems in dressing changes of burned individuals.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years,
* illiterate,
* without any mental and psychological disease and able to communicate with the assessor
* no hearing problems,
* moderate or severe burns,
* 2 days or more after burn injury,
* proliferation phase of wound healing,
* No open wound, infection or circulatory problems in the area where reflexology will be applied.
* Not having diabetes,
* not using any pre-dressing complementary medicine,
* non-pregnant,
* having no pacemaker,
* agreeing to participate in the study.

Exclusion Criteria:

* Patients who do not meet the inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-08-12 (Actual); Primary Completion 2020-03-07 (Actual); Study Completion 2020-03-07 (Actual)

PRIMARY OUTCOMES:
Pain level | 4 days
  The effect of reflexology massage and passive music on pain before burn dressing. The scale used is a scale in which the individual can score himself / herself. "0" means no pain, "10" means pain as bad as can be. In the study, patients' pain will be evaluated for 4 days before and after dressing.
Anxiety level | 4 days
  The effect of reflexology massage and passive music on anxiety before burn dressing. Anxiety of patients will be measured with Visual analog scale, State-Trait Anxiety Inventory.The Anxiety Inventory consists of two different sections and contains a total of 40 items, 20 each. Each item is scored between 1 and 4. A high score indicates that anxiety level is high. In the study, patients' anxiety will be evaluated for 4 days before and after dressing
Sleep quality | 4 days
  The effect of reflexology massage and passive music on sleep qualty before burn dressing. Sleep quality of patients will be measured by Richard-Campbell Sleep Questionnaire.Each item of the scale is evaluated between 0-100. 0-25 points indicate "very bad sleep" and 76-100 points indicate "very good sleep". The higher the scale score, the higher the sleep quality of the patient. In the study, patients' sleep will be evaluated for 4 days before and after dressing

CONTACTS AND LOCATIONS:
Locations (1):
- Ayse Kabuk, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The work is still underway and is being monitored by a committee. It is also a doctoral thesis. Necessary comments will be received and then shared.

REFERENCES:
- [Background] Molavi Vardanjani M, Masoudi Alavi N, Razavi NS, Aghajani M, Azizi-Fini E, Vaghefi SM. A randomized-controlled trial examining the effects of reflexology on anxiety of patients undergoing coronary angiography. Nurs Midwifery Stud. 2013 Sep;2(3):3-9. doi: 10.5812/nms.12167. Epub 2013 Sep 15. PMID 25414869
- [Background] Rohilla L, Agnihotri M, Trehan SK, Sharma RK, Ghai S. Effect of Music Therapy on Pain Perception, Anxiety, and Opioid Use During Dressing Change Among Patients With Burns in India: A Quasi-experimental, Cross-over Pilot Study. Ostomy Wound Manage. 2018 Oct;64(10):40-46. PMID 30312157
- [Background] Rafii F, Mohammadi-Fakhar F, Jamshidi Orak R. Effectiveness of jaw relaxation for burn dressing pain: randomized clinical trial. Pain Manag Nurs. 2014 Dec;15(4):845-53. doi: 10.1016/j.pmn.2013.11.001. Epub 2014 Apr 24. PMID 24767806